CLINICAL TRIAL: NCT03813498
Title: Health Education Based on We Media to Promote Patient Adherence to HCV Treatment: A Nationwide Online Randomized Controlled Trial
Brief Title: Hepatitis C Patient Management and Family Health Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Liver Health (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IN-CN-987-5377
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: HCV articles
- control group (Other)
  Interventions: Behavioral: general health articles

INTERVENTIONS:
Behavioral: HCV articles — The intervention group receive a targeted short article on HCV from WeChat weekly.
  Arms: intervention group
Behavioral: general health articles — The control group receive a general health article with no mention of HCV from WeChat weekly.
  Arms: control group

SUMMARY:
INTRODUCTION: Hepatitis C virus (HCV) is recognized as the leading cause of chronic liver disease worldwide. However, the screening rate and treatment rate of HCV-infected patients in China is low, which increases the burden of patients and the infection risk of their family members. WeChat, an instant messaging software, is used in a very high proportion in China. Health promotion based on WeChat public platform is a very convenient and effective way of health education. Therefore, this study plans to apply WeChat to conduct health intervention for HCV-infected patients. The objective is to explore the effect of We-media-based health promotion method on the detection rate and treatment rate of HCV-infected and their family members.

METHOD: Recruitment will be conduct in 10 hospitals in Jilin, Beijing, Henan and Anhui provinces. The subjects should be patients new diagnosed with hepatitis C at the hospital and aged 18 to 69. After signing the consent form, eligible participants were selected through the inclusion and exclusion criteria. 1000 participants will be recruited for the trial. After completing an baseline reseach by a online questionnaire, patients will be randomly assigned to receive a targeted short article on HCV weekly or a general health article with no mention of HCV. The intervention will last three months and a follow-up will be conduct at three month after the last intervention.

OUTCOMES: The primary outcome is antiviral therapy. The secondary outcomes are cognition and attitude towards hepatitis C, factors influencing antiviral therapy, time to first treatment and the compliance of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residents in the province
* Ages 18-69 (inclusive)
* Both blood anti-HCV test and HCV-RNA test is positive
* Familiar with the use of mobile phones and WeChat
* Informed consent and voluntary participation in the study

Exclusion Criteria:

* Temporary staff who come to the city to work, travel or visit relatives, or those who will be living in other cities for a long time
* Suffering from other serious diseases
* Patients with mental disorder or memory disorder
* Pregnant women or those who have a plan to prepare for pregnancy within one year
* Refuse to participate in the investigation

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Rate of antiviral therapy | 6 months after the first intervention
  The rate of antiviral therapy is equal to the number of subjects received antiviral therapy divide by the number of all subjects.

SECONDARY OUTCOMES:
Time to first treatment | 6 months after the first intervention
  This is the interval time between the first intervention and first treatment. We want to know from this outcome how long it takes the subject to receive the health intervention before starting treatment. Thus, we can analyze the relationship between intervention time and treatment behavior.
Cognition and attitude towards hepatitis C | 6 months after the first intervention
  Investigators designed a standardized questionnaire that asked questions about subjects' knowledge and attitudes toward hepatitis C. The scores of the questionnaire were used to evaluate the cognition and attitude of the subjects.
Factors influencing antiviral therapy | 6 months after the first intervention
  The investigators designed a ranking question of factors that interfered with the subjects' treatment in the questionnaire. These factors include: (1) My condition is not serious; (2) I am worried about the side effects of treatment; (3) I am afraid of being discriminated against because someone know I have the disease; (4) I have financial difficulties (or the treatment costs are too high); (5) The process of visiting a doctor is complicated. Subjects can also fill in their own ideas in the blank if they have other factors not mentioned in this questionnaire. Investigators will analyze the extent to which each factor affects a patient's treatment.
The rate of giving up treatment halfway | 6 months after the first intervention
  This rate is used to assess compliance with treatment. This rate is equal to the number of subjects who give up treatment halfway divided by the number of subjects who get treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fuqiang Cui, PhD, Study Director — Peking University; Tianshuo Zhao, Principal Investigator — Study Director; Yingsheng Shen, Principal Investigator — China Liver Health